CLINICAL TRIAL: NCT04398693
Title: Evaluation of Intestinal Microbiota Manipulation to Treat Resistant Hypertension
Acronym: VALORIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Collaborators: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, JOSE FERNANDO VILELA-MARTIN, Principal Investigator and Clinical Professor, Hospital de Base
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VALORIS
Record Dates: First submitted 2019-10-06; First posted 2020-05-21 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; Resistant Hypertension
Keywords: Microbiota; Gastrointestinal Microbiome; Hypertension; Randomized Controlled Study; Prebiotics
MeSH Terms: conditions — Hypertension | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: It shall be a double-blinded, randomized, placebo-controlled crossover study and treatment with prebiotic for 4 weeks. After a washout period of 4 weeks, the study protocol will be repeated in the other arm. Participants will receive supplementary diet based on high-amylose cornstarch, which releases large amounts of acetate and butyrate in a sachet with a powder that must be dissolved in a glass of liquid during 4 weeks (20 g 2x/day). Participants will undergo anthropometric, biochemistry and GUT microbiota assessment, before and after the end of the first phase of the crossover study. Later, when the inversion of the treatment groups occur all participants will also be subjected to the same procedures before and after the end of the second phase of the study. Afterwards, endothelial function studies, evaluating the vasodilation mediated by flow (flow-mediated dilation-FMD), and peripheral and central hemodynamics are also performed before and after the two treatment periods.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normotensive Patients (No Intervention): 40 normotensive patients with systolic BP (SBP) < 140 mmHg and diastolic BP (DBP) < 90 mmHg at the office, without the use of antihypertensive drugs and evaluated through ambulatory blood pressure monitoring (ABPM) to confirm normotension (BP < 130/80 mmHg) and the exclusion of possible masked hypertension.
- Controlled Hypertensive Patients (No Intervention): 40 controlled hypertensive patients using up to three antihypertensive drugs with SBP < 130 mmHg and DBP < 80 mmHg evaluated through 24 hours ambulatory blood pressure monitoring (ABPM).
- Resistant Hypertensive Patients (Active Comparator): The study will be double-blinded, randomized, placebo-controlled crossover Initially, 20 individuals of the resistant hypertensive group will take prebiotic for 4 weeks, while other 20 individuals this group will use placebo. After a washout period of 4 weeks, the study protocol will be repeated in the other arm.
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — It shall be a double-blinded, randomized, placebo-controlled crossover study and treatment with prebiotic for 4 weeks. After a washout period of 4 weeks, the study protocol will be repeated in the other arm. Participants will receive supplementary diet based on high-amylose cornstarch, which releases large amounts of SCFA (acetate and butyrate) in a sachet with a powder that must be dissolved in a glass of liquid to your choice, during 4 weeks (20 g 2x/day). Participants will undergo anthropometric, biochemistry and GUT microbiota assessment, before and after the end of the first phase of the crossover study. Later, when the inversion of the treatment groups occur all participants will also be subjected to the same procedures before and after the end of the second phase of the study.
  Arms: Resistant Hypertensive Patients

SUMMARY:
The gastrointestinal tract begins its colonization shortly after birth. During the first two years of life, gut microbiota is unstable and less diverse than in adulthood. Its complexity and diversity are modified by external factors that shall influence the composition of gut microbiota, especially the diet, the personal hygiene and the food cleansing, as well as the chronic use of antibiotics. Some recent evidence suggests that the microbiome may affect the likelihood of various diseases, including obesity, diabetes and cardiovascular disease. Among cardiovascular diseases, hypertension (HT) accompanied with increased cardiovascular morbidity and mortality. Hypertensive individuals may present controlled blood pressure (use of up to 03 antihypertensive drugs) or resistant without blood pressure control, even in the use of 03 or more antihypertensive drugs. Objectives: Evaluating gut microbiota of resistant hypertensive individuals, we shall compare it with those of normotensive and controlled hypertensive individuals. The resistant hypertensive ones will also receive a therapeutic intervention with prebiotics to determine if the changes in microbiota and in the production of microbiota metabolites can lower blood pressure. Methods: The study will be composed of two phases, one observational and one interventional. The observational phase will be composed of adults of both genders, aged between 40 and 70 years old, divided into three groups: normotensive, controlled hypertensive and resistant hypertensive individuals. Nutritional assessment, biochemistry and stool analysis will be performed to study the microbiota in all groups, in addition to the evaluation of peripheral and central hemodynamic parameters. The intervention phase will consist of a, randomized, double-blinded, placebo-controlled crossover study using a prebiotic formula during 04 weeks in the resistant hypertensive group. After a washout period of 4 weeks, the protocol will be repeated in the other arm. Participants will visit the clinic in 4 occasions, which shall include biochemical tests [for small chain fatty acids (SCFAs), noradrenaline, gut dysbiosis, immunomodulation] and fecal sample collection (for SCFAs and gut microbiome determination), besides the evaluation of flow-mediated dilation and peripheral and central hemodynamic parameters.

DETAILED DESCRIPTION:
The gastrointestinal tract begins its colonization shortly after the birth. During the first two years of life, microbiota is unstable and less diverse than in adulthood, when its complexity and diversity are modified. There are more than 100 trillion microorganisms hosted in the gut, mostly as phylae, Bacteroidetes and Firmicutes. These microorganisms help in various functions, and their balance is of great importance to control diseases and metabolic disorders. The lack of homeostasis of gut microbiota, results in gut dysbiosis, known by the imbalance of Firmicutes and Bacteroidetes concentration, but also with the presence of other phylae. Hypertension (HT) is characterized by blood pressure (BP) ≥ 140/90 mmHg HT can manifest itself with chronic or acute elevation of BP. Among the situations of BP chronic elevation, there is resistant hypertension (RH), defined by BP ≥ 140/90 mmHg, even with the use of three or more antihypertensive drugs in appropriate doses, preferably including a diuretic. Certain gut microbial strains may play either a pathogenic or protective role in the development hypertension. Changes in gut microbiota were observed in the hypertension with significant decrease in microbial richness, diversity and uniformity, in addition to an increased Firmicutes/Bacteroidetes ratio, characterizing intestinal dysbiosis. These changes have been accompanied by decreases in acetate and butyrate producing bacteria.

Thus, one of the mechanisms by which the gut microbiota may interfere with control of the BP is related to the production of metabolites produced by fermentation of fibers like resistant starch, known as short chain fatty acids (SCFAs). These metabolites have vasodilating property (acetate, butyrate and propionate), which may influence vascular tone. Acetate and the propionate are able to reduce the levels of BP in animal models, and that independent models of hypertension (SHR rats and Ang II), have less SCFAs producing bacteria than the normotensive controls. The SCFA butyrate, bacterial metabolic product, is produced from dietary fibers by bacteria found in lumen and hosts multiple beneficial properties for the host. Studies in animal models show that diet high in fiber and acetate supplementation correct gut dysbiosis, increase the abundance of acetate/butyrate producing bacteria and are associated with lower BP in hypertension animal model.

The spontaneously hypertensive rats prone to stroke (stroke-prone SHR) show gut dysbiosis and fecal microbiota transplant of these rats to normotensive Wistar-Kyoto rats increases the BP in normotensive rats. On the other hand, the intimate association between inflammation and chronic hypertension is well known. The control of inflammation by the sympathetic nervous system plays a central role in hypertension. Therefore, the gut receives significant sympathetic innervation, it is densely populated with a diverse microbial ecosystem, and contains immune cells that cause great impact overall inflammatory homeostasis. This influence can be demonstrated in germ-free mice subjected to the model of hypertension with infusion of Ang II. They showed mitigated inflammatory signs (smaller vascular leukocyte adhesion, smaller neutrophils and monocytes infiltration in the arterial wall), as well as smaller endothelial dysfunction and increased attenuation of the BP as a response to Ang II compared to conventionally raised mice, indicating systemic protection of inflammatory cardiovascular stress. Thus, the gut microbiota plays a key role in the immune system and can also influence the inflammatory response, by changing the endothelial function and, consequently, BP. Hypertension causes a vascular endothelium injury, triggering an inflammatory response that is accompanied with an increase in C-reactive protein, which can induce the PAI-1.

The use of Prebiotics to treat hypertension Epidemiological studies suggest that dietary components, such as fiber, may reduce the development of HT. A high fiber diet consumption increases gut microbiota populations which generate SCFAs such as acetate and butyrate. Recently, Marques et al. have shown that a high-fiber diet or supplementation with the short-chain fatty acid acetate modulated gut microbiota and prevented BP elevation and the development of cardio-renal complications in DOCA-salt hypertension rats. The authors validated these findings in hypertensive model induced by angiotensin II infusion (Ang II), showing that other SCFA, butyrate, also reduced the BP and accompanied with lower levels of inflammatory cytokines in the large bowel (data not published). Hypertensive subjects also show an abnormal gut microbiota and lower production of acetate and butyrate. Prebiotics modified diets based on high-amylose corn starches, which release large amounts of SCFAs (acetate and butyrate) into the gut and into peripheral tissues, have the ability to successfully reduce the predisposition to develop diabetes type 1 in mice and improve type II diabetes mellitus control in humans. Dietary supplements, which produce high acetate and butyrate levels, have the ability to positively intervene in gut microbiota and in chronic-metabolic diseases such as HT and diabetes, being able to be used as a new strategy to reduce the BP. Therefore, we need further investigation to assess the behavior of microbiota in controlled hypertensive and resistant hypertensive individuals and show that modulate gut microbiota can bring health benefits.

JUSTIFICATION With the high prevalence of hypertension in the globalized world and the consumption increase of industrialized foods, fast-food, ultra-processed foods and physical inactivity, there is a strong trend to the exponential growth of cardiovascular complications. Over 60 years ago, Dr. Irvine Page proposed the Mosaic Theory of Hypertension, which states that multiple factors interdigitate to blood pressure elevation. This fostered establishment of cellular, molecular, and physiological mechanisms altered in HT. However, However, how these diverse factors integrate to impair BP control remains a challenge. Furthermore, why some factors are prohypertensive in one individual and not in another, and where prohypertensive signals originate, remains an enigma. In this viewpoint, the gut microbiota can be one missing link and provide a potential unifying concept, occupying a prominent place in the mosaic theory. The latest evidence shows the involvement of the gut microbiota in BP control and its interference in HT in animal and in humans' models. Thus, addressing knowledge gaps in order to determine whether the gut microbiota is related to HT and if the change of the microbiota might help in HT treatment constitutes in an opportunity to develop new evidence to advance in this field, mainly in cases of resistant hypertension. It would be important to establish metabolites signatures and the microbiota that could be used to predict the development of HT or biomarkers for resistant hypertension. Despite great advances in drug therapy, HT continues to be the main modifiable risk factor for cardiovascular morbidity and mortality development, due to lack of BP proper control in resistant hypertension, which corresponds to about 10 to 20% of hypertensive subjects, this group is exposed to higher cardiovascular risk. Thus, this study will assess whether the gut microbiota is associated with BP levels of resistant hypertensive individuals compared to hypertensive controlled and whether the microbiota alteration with Prebiotics may help BP control and, consequently, decrease the prevalence of CVD in hypertensive patients. Additionally, this study compares the microbiota of two different global regions, Brazil and Australia, in relation to BP. Our hypothesis is that the gut microbiota and its metabolites acetate and butyrate play a role in the hypertension prevention and that medical diets ("Nutrigenomics") can be used to reduce the BP. Initially, the study will evaluate the microbiota of 3 different groups: normotensive, hypertensive controlled and resistant hypertensive individuals. In a second phase of this project, we propose the establishment of a randomized, blinded, placebo-controlled cross-over study using a prebiotic (dietary modified supplement). The use of Prebiotic is justified because it is a cheap, safe and simple therapy, constituting a new therapeutic approach that can increase BP control in resistant hypertensive patients who cannot control it with traditional drugs.

OBJECTIVES General objective The aim of this study is to evaluate the gut microbiota of resistant hypertensive patients, compared to normotensive and hypertensive ones, and also to evaluate the gut microbiota response to medical intervention (Prebiotics) in resistant hypertensive patients.

Specific objectives

* To analyze which bacteria, colonize the resistant hypertensive intestine, comparing them to the microbiota bacteria of normotensive and hypertensive controlled patients;
* To assess the patients' nutritional status studied and correlate it with their microbiota;
* To correlate metabolic-biochemistry profile (including inflammatory markers) and peripheral and central hemodynamic parameters of the patients who will be studied with the results of their microbiota evaluation;
* To carry out the intervention with the Prebiotics formula and reassess the gut microbiota after the treatment of the hypertensive controlled and the resistant hypertensive group.
* To compare the microbiota of normotensive, hypertensive controlled and resistant hypertensive of Brazilian population studied with Australians.

MATERIALS AND METHODS The study shall be divided into two phases. The first phase will be a descriptive, observational cross-sectional study. The collection of material shall be carried out at the Hypertension Clinic of State Medical School at São José do Rio Preto (FAMERP), with the aim of evaluating the gut microbiota of normotensive, hypertensive controlled and resistant hypertensive patients. The second study will be a randomized, blinded, placebo-controlled crossover study, using prebiotics in resistant hypertensive patients during two periods of 4 weeks with a wash-out interval of 4 weeks.

Characteristics of the participants

Patients who are being monitored will be assessed at the Hypertension Clinic. The study will consist of 3 groups of participants:

1. 40 normotensive patients with systolic BP (SBP) < 140 mmHg and diastolic BP (DBP) < 90 mmHg at the office, without the use of antihypertensive drugs and evaluated through ambulatory blood pressure monitoring (ABPM) to confirm normotension (BP < 130/80 mmHg) and the exclusion of possible masked hypertension.
2. 40 controlled hypertensive patients using up to three antihypertensive drugs with SBP < 130 mmHg and DBP < 80 mmHg evaluated through ambulatory blood pressure monitoring (ABPM).
3. 40 resistant hypertensive patients defined by an uncontrolled BP in doctor's office (≥ 140/90 mmHg), despite the use of three or more antihypertensive drugs in appropriate doses, including preferably a diuretic, or the use of four or more drugs with blood pressure control. Patients will also be evaluated by the ABPM, which should present in SBP ≥130 mmHg and DBP ≥ 80 mmHg to be considered resistant hypertensive, otherwise they will be classified as controlled hypertensive. Resistant hypertension will be defined after the exclusion of causes of pseudo-resistance, i.e., inaccurate blood pressure measurement, white coat effect, non-therapeutic adherence, the use of drugs that can increase BP and secondary causes of arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Be normotensive, controlled hypertensive or resistant hypertensive.
* Body Mass Index (BMI) < 35 kg/m 2 .
* If diabetic, glycated hemoglobin must be ≤ 9.0%.
* Agree and sign the Free Informed Consent Form (FICF).

Exclusion Criteria:

* BMI ≥ 35 kg/m 2 ;
* Urinary Sodium ≥ 200mEq/L in 24-hour urine;
* Bariatric Surgery;
* Recent use of antibiotics or probiotics (<3 months);
* Prior Cardiovascular Disease: Acute Myocardial Infarction, Stroke, Heart Failure, Angina Pectoris, Peripheral Arterial Insufficiency;
* Chronic kidney disease (glomerular filtration rate (GFR) < 30 mL/min/m 2 );
* Chronic Disease limiting participation at the study or life expectancy (e.g.: cancer, among others);
* Gastrointestinal diseases (including inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis or other disabsortive disease)
* Pregnant or having the intension of become pregnant in the next two years;
* Participation in any other clinical studies in the past six months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure | 12 weeks
  This study will provide a background for the use of a new strategy to lower the BP. The study primary outcome will be to observe the lowering of blood pressure.

SECONDARY OUTCOMES:
Change of inflammatory activity | 12 weeks
  Changes in inflammatory cytokines and/or in immune cells
Microbiota modulation | 12 weeks
  Changes in the microbiota modulation dietary supplement intake evaluating the richness, uniformity and microbial diversity of gut microbiota. Moreover, it will be evaluated Firmicutes/Bacteroidetes ratio considered a signature of gut dysbiosis.

CONTACTS AND LOCATIONS:
Overall Officials: José F Vilela-Martin, MD PhD FAHA, Principal Investigator — State Medical School at São José do Rio Preto (FAMERP), São Paulo, Brazil; Francine Z Marques, PhD, Principal Investigator — School of Biological Sciences, Faculty of Science, Monash University, Melbourne, VIC, Australia
Locations (1):
- State Medical School at São José do Rio Preto (FAMERP), São Paulo, Brazil, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No